CLINICAL TRIAL: NCT00001778
Title: Immuno-Virological Evaluation of Human T Cell Leukemia Virus Type-1 Associated Myelopathy (HAM/TSP)
Brief Title: Evaluation of Patients With HAM/TSP
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980047; 98-N-0047
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12-30

CONDITIONS: HTLV-I Infection; Tropical Spastic Paraparesis
Keywords: Immune Response; Sero-Indeterminant; Transmission; HTLV-1; HTLV-1 Associated Myelopathy; Natural History; HTLV-I; HAM/TSP
MeSH Terms: conditions — HTLV-I Infections; Paraparesis, Tropical Spastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers: At least 18 years old and have no history of any medical illness that may confound study results or make participation in this protocol impossible
- individuals seropositive for HTLV: Positive HTLV-1 ELISA followed by a positive Western Blot
- individuals with indeterminate HTLV sero-status: Positive HTLV ELISA but a Western Blot that only partially fulfills criteria

SUMMARY:
Objective:

Human T-lymphotropic virus type-I-associated myelopathy / tropical spastic paraparesis (HAM/TSP) is a rare neurologic disorder that affects less than 5% of patients infected with the HTLV-I virus. The purpose of this protocol is to study the natural history of HAM/TSP by monitoring clinical progression of patients longitudinally. Additionally, we will attempt to define the virological and immunological changes of HAM/TSP.

Study Population:

Patients with HAM/TSP who fulfill World Health Organization diagnostic criteria are eligible to participate in this protocol. Asymptomatic seropositive individuals and individuals with indeterminate HTLV-1 serology are also eligible to participate.

Design and Outcome Measures:

A longitudinal assessment of clinical, virological and immunological progression in HAM/TSP will be accomplished through periodic testing and evaluation. Asymptomatic seropositive individuals, those with seroindeterminate HTLV-I serology and normal volunteers may serve as controls. Longitudinal standardized neurological examinations will be performed. Longitudinal samples of serum, plasma, and lymphocytes may be obtained from participants. Lumbar punctures may be performed on all participants. These samples will be used virological and immunological assays. A focus is on the relationships between the characteristics of viral infection, the immune response, and the genetic makeup.

DETAILED DESCRIPTION:
Objective

Human T lymphotropic virus type 1 (HTLV-1) was first discovered in the search for retroviruses causing cancer in 1981. Shortly afterwards, HTLV-2 was also isolated. Although HTLV-1 and HTLV-2 share similar genome structure, routes of transmission, and replication pattern, they differ in epidemiology and disease associations. Human T-lymphotropic virus type-I-associated myelopathy / tropical spastic paraparesis (HAM/TSP) is a rare neurologic disorder that affects less than 5% of patients infected with the HTLV-I virus. Recently, a large body of literature supports other inflammatory manifestations, some neurological such as myositis, due to HTLV-1 infection. Studies of HLTV-2 clinical manifestations have largely been confounded by concomitant HIV-1 infection or IV drug abuse making the establishment of clear relationship with other manifestations such as neurological disease difficult. Most patients infected with HTLV remain asymptomatic throughout their lifetime. The purpose of this protocol is to study the natural history of HTLV infection by monitoring participants longitudinally. Additionally, we will attempt to define the virological and immunological changes of these viral infections. In addition, this protocol may be used to screen for other VIS protocols.

Study Population

Individuals sero-positive for HTLV, individuals with indeterminate HTLV sero-status, and healthy volunteers are eligible to participate in this protocol. Some individuals sero-positive for HTLV may have associated diseases including but not limited to HTLV-1 associated myelopathy/tropical spastic paraparesis (HAM/TSP) and HTLV associated inflammatory disorders.

Design & Outcome Measures

A longitudinal assessment of clinical, virological and immunological progression in HTLV related disease will be accomplished through periodic testing and evaluation. Asymptomatic seropositive individuals, those with sero-indeterminate HTLV serology and healthy volunteers may serve as controls. Longitudinal standardized neurological examinations will be performed. Longitudinal samples of serum, plasma, and lymphocytes may be obtained from participants. Lumbar punctures may be performed on all participants. These samples will be used for virological and immunological assays. A focus is on the relationships between the characteristics of viral infection, the immune response, and the genetic makeup.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants that meet one of the following criteria:

* Test positive for HTLV infection (positive HTLV-1 ELISA followed by a positive Western blot)
* Positive HTLV ELISA but a Western Blot that only partially fulfills the above criteria (seroindeterminate)
* Have a family member/significant other who is HTLV positive, and may have been exposed to the virus
* Healthy volunteer AND
* Willingness to participate in the protocol evaluations and procedures.

EXCLUSION CRITERIA:

* Unwillingness or inability to participate in the protocol evaluations and procedures.
* The presence of any medical, social, or psychiatric conditions that in the opinion of the investigator may affect the safety of the patients or compliance with the protocol.
* Patients/healthy volunteers under the age of 18 are excluded.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals sero-positive for HTLV, individuals with indeterminate HTLV sero-status, and healthy volunteers are eligible to participate in this protocol. Some individuals sero-positive for HTLV may have associated diseases including but not limited to HTLV-1 associated myelopathy/tropical spastic paraparesis (HAM/TSP) and HTLV associated inflammatory myositis.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 1998-04-06 (Actual)

PRIMARY OUTCOMES:
To characterize the baseline features of patients with HTLV infection with regards to clinical features, imaging studies, immunological markers, and viral studies. | each study visit
  To characterize the baseline features of patients with HTLV infection with regards to clinical features, imaging studies, immunological markers, and viral studies.

SECONDARY OUTCOMES:
Change in proviral load | each study visit
  Change proviral load

CONTACTS AND LOCATIONS:
Overall Officials: Steven Jacobson, Ph.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gessain A, Barin F, Vernant JC, Gout O, Maurs L, Calender A, de The G. Antibodies to human T-lymphotropic virus type-I in patients with tropical spastic paraparesis. Lancet. 1985 Aug 24;2(8452):407-10. doi: 10.1016/s0140-6736(85)92734-5. PMID 2863442
- [Background] Osame M, Matsumoto M, Usuku K, Izumo S, Ijichi N, Amitani H, Tara M, Igata A. Chronic progressive myelopathy associated with elevated antibodies to human T-lymphotropic virus type I and adult T-cell leukemialike cells. Ann Neurol. 1987 Feb;21(2):117-22. doi: 10.1002/ana.410210203. PMID 2881513
- [Background] Iwasaki Y. Pathology of chronic myelopathy associated with HTLV-I infection (HAM/TSP). J Neurol Sci. 1990 Apr;96(1):103-23. doi: 10.1016/0022-510x(90)90060-z. PMID 2351985
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1998-N-0047.html